CLINICAL TRIAL: NCT02750618
Title: An Open-Label, Phase 2 Study to Assess the Safety, Pharmacodynamics, and Efficacy of KRN23 in Children From 1 to 4 Years Old With X-linked Hypophosphatemia (XLH)
Brief Title: Study of the Safety, Pharmacodynamics (PD) and Efficacy of KRN23 in Children From 1 to 4 Years Old With X-linked Hypophosphatemia (XLH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX023-CL205
Expanded Access: NCT03775187 (Available)
Record Dates: First submitted 2015-12-06; First posted 2016-04-25 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: X-Linked Hypophosphatemia
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Burosumab Q2W (Experimental): Burosumab subcutaneous (SC) injections every 2 weeks (Q2W) for a total of 160 weeks.
  Interventions: Biological: Burosumab

INTERVENTIONS:
Biological: Burosumab — solution for subcutaneous injection
  Other Names: KRN23; Crysvita®; UX023

SUMMARY:
The primary objectives of the study are to:

* Establish the safety profile of KRN23 for the treatment of XLH in children between 1 and 4 years old
* Determine the PD effects of KRN23 treatment on serum phosphorus and other PD markers that reflect the status of phosphate homeostasis in children between 1 and 4 years old with XLH

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥1 year and <5 years
2. Diagnosis of XLH supported by ONE or more of the following

   * Confirmed phosphate regulating gene with homology to endopeptidases located on the X chromosome (PHEX) mutation in the patient or a directly related family member with appropriate X-linked inheritance
   * Serum fibroblast growth factor 23 (FGF23) level > 30 pg/mL by Kainos assay
3. Biochemical findings associated with XLH including:

   * Serum phosphorus < 3.0 mg/dL (0.97 mmol/L)
   * Serum creatinine within age-adjusted normal range
4. Radiographic evidence of rickets
5. Willing to provide access to prior medical records for the collection of historical growth, biochemical, and radiographic data and disease history
6. Provide written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures
7. Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule, and comply with the assessments

Exclusion Criteria:

1. Unwilling to stop treatment with oral phosphate and/or pharmacologic vitamin D metabolite or analog (e.g. calcitriol, alfacalcidol) during the screening period and for the duration of the study
2. Presence of nephrocalcinosis on renal ultrasound grade 4 based on the following scale: 0 = Normal, 1 = Faint hyperechogenic rim around the medullary pyramids, 2 = More intense echogenic rim with echoes faintly filling the entire pyramid, 3 = Uniformly intense echoes throughout the pyramid, 4 = Stone formation: solitary focus of echoes at the tip of the pyramid
3. Planned or recommended orthopedic surgery including staples, 8-plates or osteotomy, within the clinical trial period
4. Hypocalcemia or hypercalcemia, defined as serum calcium levels outside the age-adjusted normal limits
5. Presence or history of any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study
6. Presence of a concurrent disease or condition that would interfere with study participation or affect safety
7. History of recurrent infection or predisposition to infection, or of known immunodeficiency
8. Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (3):
- United States (3):
  - Yale University School of Medicine, New Haven, Connecticut
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Shriners Hospital for Children, St Louis, Missouri

REFERENCES:
- [Derived] Mao M, Carpenter TO, Whyte MP, Skrinar A, Chen CY, San Martin J, Rogol AD. Growth Curves for Children with X-linked Hypophosphatemia. J Clin Endocrinol Metab. 2020 Oct 1;105(10):3243-9. doi: 10.1210/clinem/dgaa495. PMID 32721016
- [Derived] Whyte MP, Carpenter TO, Gottesman GS, Mao M, Skrinar A, San Martin J, Imel EA. Efficacy and safety of burosumab in children aged 1-4 years with X-linked hypophosphataemia: a multicentre, open-label, phase 2 trial. Lancet Diabetes Endocrinol. 2019 Mar;7(3):189-199. doi: 10.1016/S2213-8587(18)30338-3. Epub 2019 Jan 9. PMID 30638856

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled pediatric participants between 1 and 4 years old, inclusive, with clinical findings consistent with XLH including hypophosphatemia and radiographic evidence of rickets, and a confirmed PHEX mutation or variant of uncertain significance.
Period: Overall Study
Arm/Group | Burosumab Q2W
Started | 13
Completed Week 40 | 13
Completed Week 64 | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Burosumab Q2W: Burosumab SC injections Q2W for a total of 160 weeks.
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.94 (1.146)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
  Black or African American | 1
Serum Phosphorus [Mean (Standard Deviation); unit: mg/dL] | 2.51 (0.284)
Rickets Severity Score (RSS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The RSS system is a 10-point radiographic scoring method that was developed to assess the severity of nutritional rickets in the wrists and knees based on the degree of metaphyseal fraying, cupping, and the proportion of the growth plate affected. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points and the minimum score is 0, with a total possible score of 4 points for the wrists and 6 points for the knees. Higher scores indicate greater rickets severity.
  units on a scale | 2.92 (1.367)
Recumbent length/Standing height [Mean (Standard Deviation); unit: cm] — Growth is measured by recumbent length for subjects < 2 years of age or those unable or unwilling to stand for the measurement.
  cm | 89.15 (7.597)
Recumbent length/Standing height (Z score) [Mean (Standard Deviation); unit: Z score] — Recumbent length/Standing height z scores are measures of height adjusted for a child's age and sex. The Z-score indicates the number of standard deviations away from a reference population (from the Centers for Disease Control [CDC] growth charts) in the same age range and with the same sex. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome.
  Z score | -1.378 (1.1947)
Recumbent length/Standing height (percentile) [Mean (Standard Deviation); unit: percentile] | 18.044 (25.2644)
Serum Alkaline Phosphatase (ALP) [Mean (Standard Deviation); unit: U/L] | 548.5 (193.80)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 40 in Serum Phosphorus
Description: The Generalized Estimation Equation (GEE) model includes the change from baseline as the dependent variable, time as the categorical variable and adjusted for baseline measurement, with exchangeable covariance structure.
Time Frame: Baseline, Week 40
Population: Pharmacokinetic/Pharmacodynamic (PK/PD) Analysis Set: all participants who received at least one dose of study drug and had evaluable blood samples.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
mg/dL | 0.96 (0.117)
Statistical Analysis 1: Comparison: Burosumab Q2W; Test type: Superiority; p < 0.0001, GEE model; Least Squares Mean Difference = 0.96, 95% CI 2-sided [0.73 to 1.19]

2. Primary Outcome: Number of Participants With Adverse Events (AEs), Treatment Emergent AEs (TEAEs), Serious TEAEs, and TEAEs Leading to Discontinuation
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug, whether or not considered drug related. A serious AE was defined as an AE that at any dose, in the view of either the Investigator or Sponsor, results in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or disability, a congenital anomaly/birth defect, or other important medical events (according to the investigator). An AE was considered a TEAE if it occurred on or after the first dose and was not present prior to the first dose, or it was present prior to the first dose but increased in severity during the study. Events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0: grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life-threatening), grade 5 (death).
Time Frame: From first dose of study drug through the end of the study (Week 160). Maximum duration of exposure to study drug was 160 weeks.
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
Participants
  Adverse Event Starting during Screening Period | 5
  TEAEs | 13
  Related TEAEs | 5
  Serious TEAEs | 1
  Serious Related TEAEs | 0
  Grade 3 or 4 TEAE | 2
  TEAE Leading to Study Discontinuation | 0
  TEAE Leading to Treatment Discontinuation | 0
  TEAE Leading to Death | 0

3. Secondary Outcome: Radiographic Global Impression of Change (RGI-C) Score at Week 40
Description: Changes in the severity of rickets and bowing were assessed centrally by three independent pediatric radiologists contracted by a central imaging facility using a disease specific qualitative RGI-C scoring system. The RGI-C is a seven point ordinal scale with possible values: +3 = very much better (complete or near complete healing of rickets), +2 = much better (substantial healing of rickets), +1 = minimally better (i.e., minimal healing of rickets), 0 = unchanged, -1 = minimally worse (minimal worsening of rickets), -2 = much worse (moderate worsening of rickets), -3 = very much worse (severe worsening of rickets). The Analysis of Covariance (ANCOVA) model includes the RGI-C score as the dependent variable, age and RSS at baseline as covariates.
Time Frame: Week 40
Population: Efficacy Analysis Set: all participants who received at least one dose of study drug and had at least one post-study drug measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
units on a scale | 2.21 (0.071)
Statistical Analysis 1: Comparison: Burosumab Q2W; Test type: Superiority; p < 0.0001, GEE model; Difference in LS Means = 2.21, 95% CI 2-sided [2.07 to 2.35]

4. Secondary Outcome: RGI-C Score at Week 64
Description: Changes in the severity of rickets and bowing were assessed centrally by three independent pediatric radiologists contracted by a central imaging facility using a disease specific qualitative RGI-C scoring system. The RGI-C is a seven point ordinal scale with possible values: +3 = very much better (complete or near complete healing of rickets), +2 = much better (substantial healing of rickets), +1 = minimally better (i.e., minimal healing of rickets), 0 = unchanged, -1 = minimally worse (minimal worsening of rickets), -2 = much worse (moderate worsening of rickets), -3 = very much worse (severe worsening of rickets). The GEE model includes the RGI-C score as the dependent variable, visit as a factor, age and RSS at baseline as covariates, with exchangeable covariance structure.
Time Frame: Week 64
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
units on a scale | 2.23 (0.111)
Statistical Analysis 1: Comparison: Burosumab Q2W; The GEE model includes the RGI-C score as the dependent variable, visit as a factor, age and RSS at baseline as covariates, with exchangeable covariance structure. The least squares (LS) mean, standard error (SE), 95% confidence interval (CI) and 2-sided p-value are from the GEE model; Test type: Superiority; p < 0.0001, GEE model; Difference in LS Means = 2.23, 95% CI 2-sided [2.01 to 2.45]

5. Secondary Outcome: Change From Baseline in Rickets at Week 40 as Assessed by the RSS Total Score
Description: The RSS system is a 10-point radiographic scoring method that was developed to assess the severity of nutritional rickets in the wrists and knees based on the degree of metaphyseal fraying, cupping, and the proportion of the growth plate affected. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points and the minimum score is 0, with a total possible score of 4 points for the wrists and 6 points for the knees. Higher scores indicate greater rickets severity.The ANCOVA model includes the RGI-C score as the dependent variable, age and RSS at baseline as covariates.
Time Frame: Baseline, Week 40
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
units on a scale | -1.75 (0.116)
Statistical Analysis 1: Comparison: Burosumab Q2W; Test type: Superiority; p < 0.0001, GEE model; Difference in LS Means = -1.75, 95% CI 2-sided [-1.98 to -1.53]

6. Secondary Outcome: Change From Baseline in Rickets at Week 64 as Assessed by the RSS Total Score
Description: The RSS system is a 10-point radiographic scoring method that was developed to assess the severity of nutritional rickets in the wrists and knees based on the degree of metaphyseal fraying, cupping, and the proportion of the growth plate affected. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points, with a total possible score of 4 points for the wrists and 6 points for the knees. Higher scores indicate greater rickets severity. The GEE model includes the change from baseline in RSS as the dependent variable, visit as a factor, age and RSS at baseline as covariates, with exchangeable covariance structure.
Time Frame: Baseline, Week 64
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
units on a scale | -2.02 (0.115)
Statistical Analysis 1: Comparison: Burosumab Q2W; Test type: Superiority; p < 0.0001, GEE model — The GEE model includes the change from baseline in RSS as the dependent variable, visit as a factor, age and RSS at baseline as covariates, with exchangeable covariance structure; Difference in LS Means = -2.02, 95% CI 2-sided [-2.25 to -1.80]

7. Secondary Outcome: RGI-C Lower Limb Deformity Score at Week 40
Description: Changes in the severity of lower extremity skeletal abnormalities were assessed centrally by three independent pediatric radiologists contracted by a central imaging facility using a disease specific qualitative RGI-C scoring system. The RGI-C is a seven point ordinal scale with possible values: +3 = very much better (complete or near complete healing of rickets), +2 = much better (substantial healing of rickets), +1 = minimally better (i.e., minimal healing of rickets), 0 = unchanged, -1 = minimally worse (minimal worsening of rickets), -2 = much worse (moderate worsening of rickets), -3 = very much worse (severe worsening of rickets). The ANCOVA model includes the RGI-C score as the dependent variable, age and RSS at baseline as covariates.
Time Frame: Week 40
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
units on a scale | 1.21 (0.155)
Statistical Analysis 1: Comparison: Burosumab Q2W; Test type: Superiority; p < 0.0001, GEE model; Difference in LS Means = 1.21, 95% CI 2-sided [0.90 to 1.51]

8. Secondary Outcome: RGI-C Lower Limb Deformity Score at Week 64
Description: Changes in the severity of lower extremity skeletal abnormalities were assessed centrally by three independent pediatric radiologists contracted by a central imaging facility using a disease specific qualitative RGI-C scoring system. The RGI-C is a seven point ordinal scale with possible values: +3 = very much better (complete or near complete healing of rickets), +2 = much better (substantial healing of rickets), +1 = minimally better (i.e., minimal healing of rickets), 0 = unchanged, -1 = minimally worse (minimal worsening of rickets), -2 = much worse (moderate worsening of rickets), -3 = very much worse (severe worsening of rickets). The GEE model includes the RGI-C score as the dependent variable, visit as a factor, age and RSS at baseline as covariates, with exchangeable covariance structure.
Time Frame: Week 64
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
units on a scale | 1.51 (0.123)
Statistical Analysis 1: Comparison: Burosumab Q2W; Test type: Superiority; p < 0.0001, GEE — The GEE model includes the RGI-C score as the dependent variable, visit as a factor, age and RSS at baseline as covariates, with exchangeable covariance structure. The LS Mean, SE, 95% CI and 2-sided p-value are from the GEE model; Difference in LS Means = 1.51, 95% CI 2-sided [1.27 to 1.76]

9. Secondary Outcome: Change From Baseline Over Time in Recumbent Length/Standing Height
Time Frame: Baseline, Weeks 12, 24, 40, 64, 88, 112, 136, 160
Population: Efficacy Analysis Set: all participants who received at least one dose of study drug and had at least one post-study drug measurement at given time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
cm
  Week 12 | 1.44 (2.009)
  Week 24 | 2.52 (1.518)
  Week 40 | 4.29 (2.451)
  Week 64 | 7.22 (3.157)
  Week 88 | 10.30 (3.400)
  Week 112 | 13.25 (3.724)
  Week 136: number analyzed (Participants) | 11
  Week 136 | 15.41 (3.699)
  Week 160: number analyzed (Participants) | 12
  Week 160 | 18.96 (4.206)

10. Secondary Outcome: Change From Baseline Over Time in Recumbent Length/Standing Height as Assessed by Height-for-Age Z-Scores
Description: Recumbent length/Standing height z scores are measures of height adjusted for a child's age and sex. The Z-score indicates the number of standard deviations away from a reference population (from the CDC growth charts) in the same age range and with the same sex. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome.
Time Frame: Baseline, Weeks 12, 24, 40, 64, 88, 112, 136, 160
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
Z score
  Week 12 | -0.082 (0.4964)
  Week 24 | -0.208 (0.4540)
  Week 40 | -0.276 (0.6647)
  Week 64 | -0.264 (0.8755)
  Week 88 | -0.212 (0.9115)
  Week 112 | -0.174 (0.9273)
  Week 136: number analyzed (Participants) | 11
  Week 136 | -0.321 (0.9123)
  Week 160: number analyzed (Participants) | 12
  Week 160 | -0.172 (0.9048)

11. Secondary Outcome: Change From Baseline Over Time in Recumbent Length/Standing Height as Assessed by Percentiles
Time Frame: Baseline, Weeks 12, 24, 40, 64, 88, 112, 136, 160
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentiles
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
percentiles
  Week 12 | -0.006 (11.6149)
  Week 24 | -4.940 (13.1323)
  Week 40 | -5.283 (20.1675)
  Week 64 | -4.980 (23.4412)
  Week 88 | -4.155 (23.9126)
  Week 112 | -3.000 (24.7569)
  Week 136: number analyzed (Participants) | 11
  Week 136 | -7.026 (24.8583)
  Week 160: number analyzed (Participants) | 12
  Week 160 | -3.628 (25.5113)

12. Secondary Outcome: Change From Baseline Over Time in Serum Alkaline Phosphatase (ALP)
Description: The GEE model includes the change from baseline as the dependent variable, time as the categorical variable and adjusted for baseline measurement, with exchangeable covariance structure.
Time Frame: Baseline, Weeks 4, 12, 20, 40, 48, 56, 64, 76, 88, 100, 112, 124, 136, 148, 160
Population: PK/PD Analysis Set: all participants who received at least one dose of study drug and had evaluable blood samples at given time point.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
U/L
  Week 4 | -82.91 (23.348)
  Week 12 | -83.84 (45.263)
  Week 20 | -161.38 (12.924)
  Week 40 | -214.99 (13.628)
  Week 48: number analyzed (Participants) | 12
  Week 48 | -226.58 (11.491)
  Week 56 | -216.45 (16.165)
  Week 64 | -216.76 (12.705)
  Week 76 | -231.22 (15.964)
  Week 88: number analyzed (Participants) | 12
  Week 88 | -237.78 (12.837)
  Week 100 | -218.14 (15.340)
  Week 112 | -233.91 (11.098)
  Week 124: number analyzed (Participants) | 12
  Week 124 | -252.22 (8.312)
  Week 136: number analyzed (Participants) | 12
  Week 136 | -267.89 (13.124)
  Week 148: number analyzed (Participants) | 12
  Week 148 | -248.05 (12.653)
  Week 160: number analyzed (Participants) | 12
  Week 160 | -248.47 (10.990)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 4; Test type: Superiority; p = 0.0004, GEE model; Difference in LS Means = -82.91, 95% CI 2-sided [-128.68 to -37.15]
Statistical Analysis 2: Comparison: Burosumab Q2W; Week 12; Test type: Superiority; p = 0.0640, GEE model; Difference in LS Means = -83.84, 95% CI 2-sided [-172.55 to 4.88]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 20; Test type: Superiority; p < 0.0001, GEE model; Difference in LS Means = -161.38, 95% CI 2-sided [-186.70 to -136.05]
Statistical Analysis 4: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, GEE model; Difference in LS Means = -214.99, 95% CI 2-sided [-241.70 to -188.28]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 48; Test type: Superiority; p < 0.0001, GEE model; Difference in LS Means = -226.58, 95% CI 2-sided [-249.11 to -204.06]
Statistical Analysis 6: Comparison: Burosumab Q2W; Week 56; Test type: Superiority; p < 0.0001, GEE model; Difference in LS Means = -216.45, 95% CI 2-sided [-248.13 to -184.77]
Statistical Analysis 7: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model; Difference in LS Means = -216.76, 95% CI 2-sided [-241.66 to -191.86]
Statistical Analysis 8: Comparison: Burosumab Q2W; Week 76; Test type: Superiority; p < 0.0001, GEE; LS Mean = -231.22, 95% CI 2-sided [-262.51 to -199.93]
Statistical Analysis 9: Comparison: Burosumab Q2W; Week 88; Test type: Superiority; p < 0.0001, GEE; LS Mean = -237.78, 95% CI 2-sided [-262.94 to -212.62]
Statistical Analysis 10: Comparison: Burosumab Q2W; Week 100; Test type: Superiority; p < 0.0001, GEE; LS Mean = -218.14, 95% CI 2-sided [-248.21 to -188.08]
Statistical Analysis 11: Comparison: Burosumab Q2W; Week 112; Test type: Superiority; p < 0.0001, GEE; LS Mean = -233.91, 95% CI 2-sided [-255.66 to -212.16]
Statistical Analysis 12: Comparison: Burosumab Q2W; Week 124; Test type: Superiority; p < 0.0001, GEE; LS Mean = -252.22, 95% CI 2-sided [-268.51 to -235.93]
Statistical Analysis 13: Comparison: Burosumab Q2W; Week 136; Test type: Superiority; p < 0.0001, GEE; LS Mean = -267.89, 95% CI 2-sided [-293.61 to -242.16]
Statistical Analysis 14: Comparison: Burosumab Q2W; Week 148; Test type: Superiority; p < 0.0001, GEE; LS Mean = -248.05, 95% CI 2-sided [-272.85 to -223.25]
Statistical Analysis 15: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE; LS Mean = -248.47, 95% CI 2-sided [-270.01 to -226.93]

13. Secondary Outcome: Percent Change From Baseline Over Time in Serum ALP
Time Frame: Baseline, Weeks 4, 12, 20, 40, 48, 56, 64, 76, 88, 100, 112, 124, 136, 148, 160
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Burosumab Q2W
Number analyzed (Participants) | 13
percent change
  Week 4 | -12.47 (16.620)
  Week 12 | -5.00 (60.124)
  Week 20 | -24.76 (18.883)
  Week 40 | -36.25 (12.787)
  Week 48 | -37.29 (13.936)
  Week 56 | -35.80 (16.568)
  Week 64 | -35.95 (14.851)
  Week 76 | -38.36 (15.621)
  Week 88: number analyzed (Participants) | 12
  Week 88 | -39.08 (12.987)
  Week 100 | -37.42 (12.466)
  Week 112 | -39.05 (13.808)
  Week 124: number analyzed (Participants) | 12
  Week 124 | -43.11 (12.493)
  Week 136: number analyzed (Participants) | 12
  Week 136 | -47.01 (11.752)
  Week 148: number analyzed (Participants) | 12
  Week 148 | -43.47 (11.321)
  Week 160: number analyzed (Participants) | 12
  Week 160 | -42.35 (13.574)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of the study (at Week 160). Maximum duration of exposure to study drug was 160 weeks.
Arm/Group | Burosumab Q2W
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Burosumab Q2W (N=13)
Tooth Abscess (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Burosumab Q2W (N=13)
Skull Malformation (Congenital, familial and genetic disorders) | 1
Syringomyelia (Congenital, familial and genetic disorders) | 1
Deafness Unilateral (Ear and labyrinth disorders) | 1
Ear Haemorrhage (Ear and labyrinth disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 4
Excessive Cerumen Production (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Motion Sickness (Ear and labyrinth disorders) | 1
Otorrhoea (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Ocular Hyperaemia (Eye disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 5
Aphthous Ulcer (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dental Caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Epigastric Discomfort (Gastrointestinal disorders) | 1
Gingival Blister (Gastrointestinal disorders) | 1
Gingival Erythema (Gastrointestinal disorders) | 1
Gingival Pain (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Loose Tooth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral Pain (Gastrointestinal disorders) | 4
Post-Tussive Vomiting (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Teething (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 7
Vomiting Projectile (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Injection Site Bruising (General disorders) | 1
Injection Site Erythema (General disorders) | 2
Injection Site Pain (General disorders) | 1
Injection Site Pruritus (General disorders) | 2
Injection Site Reaction (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 11
Vaccination Site Reaction (General disorders) | 1
Food Allergy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 3
Atypical Pneumonia (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Croup Infectious (Infections and infestations) | 1
Ear Infection (Infections and infestations) | 6
Enterobiasis (Infections and infestations) | 1
Eye Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal Viral Infection (Infections and infestations) | 1
Genital Candidiasis (Infections and infestations) | 1
Gingival Abscess (Infections and infestations) | 1
Hand-Foot-And-Mouth Disease (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Impetigo (Infections and infestations) | 2
Influenza (Infections and infestations) | 3
Molluscum Contagiosum (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Otitis Media (Infections and infestations) | 1
Pharyngitis Streptococcal (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Tooth Abscess (Infections and infestations) | 10
Upper Respiratory Tract Infection (Infections and infestations) | 9
Urinary Tract Infection (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 2
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3
Arthropod Bite (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 4
Laceration (Injury, poisoning and procedural complications) | 1
Lip Injury (Injury, poisoning and procedural complications) | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 4
Tooth Fracture (Injury, poisoning and procedural complications) | 1
Tooth Injury (Injury, poisoning and procedural complications) | 1
Traumatic Tooth Displacement (Injury, poisoning and procedural complications) | 1
Amylase Increased (Investigations) | 2
Blood 25-Hydroxycholecalciferol Decreased (Investigations) | 1
Blood Parathyroid Hormone Increased (Investigations) | 1
Blood Phosphorus Decreased (Investigations) | 1
Heart Rate Abnormal (Investigations) | 1
Lipase Increased (Investigations) | 1
Vitamin D Decreased (Investigations) | 2
White Blood Cell Count Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Increased Appetite (Metabolism and nutrition disorders) | 1
Polydipsia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 3
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1
Knee Deformity (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Hypersomnia (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Periodic Limb Movement Disorder (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Penile Erythema (Reproductive system and breast disorders) | 1
Penile Pain (Reproductive system and breast disorders) | 1
Adenoidal Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Throat Clearing (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 8
Nasal Discharge Discolouration (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Rash Papular (Skin and subcutaneous tissue disorders) | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4
Urticaria Papular (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT02750618/Prot_002.pdf
  • Statistical Analysis Plan (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT02750618/SAP_001.pdf